CLINICAL TRIAL: NCT05404100
Title: Effects of Aortic Valve Replacement on Myocardial T1 Values in Severe Aortic Valve Stenosis
Acronym: FIBROTIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cardiovascular Academy (DCA) (Unknown); Eva og Henry Frænkels Mindefond (Other); Snedkermester Sophus Jacobsen and hustru Astrid Jacobsens Foundation (Other)
Responsible Party: Principal Investigator, Katrine Aagaard Myhr, Principtal Investigator, Rigshospitalet, Denmark
Other Study IDs: H-20029458
Record Dates: First submitted 2022-05-25; First posted 2022-06-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Replacement; Myocardial Fibrosis; Cardiac Magnetic Resonance; T1 Mapping
Keywords: Aortic Valve Stenosis; Aortic Valve Replacement; Myocardial Fibrosis; Cardiac Magnetic Resonance; T1 mapping
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe aortic valve stenosis: Patients with severe AS planned to undergo AVR, either as surgical aortic valve replacement (SAVR) or transcatheter aortic valve replacement (TAVR).
  Interventions: Procedure: Aortic valve replacement

INTERVENTIONS:
Procedure: Aortic valve replacement — SAVR or TAVR

SUMMARY:
Background: Severe aortic valve stenosis (AS) is the commonest valve disease. Aortic valve replacement (AVR) is primarily indicated when symptoms occur and/or when there is a drop in left ventricular ejection fraction. However, irreversible myocardial damage, such as replacement fibrosis, leads to increased morbidity and mortality despite treatment. Improved patient selection and timely treatment is thus warranted. T1 mapping, a non-invasive method to quantify myocardial fibrosis by cardiac magnetic resonance (CMR), could be a marker to guide treatment.

Aims: To investigate the change of myocardial fibrosis* in AS patients following AVR and if these changes are associated with disease and/or procedural characteristics.

Methods: This is an observational clinical trial. Approximately 60 patients with severe AS planned to undergo AVR (either surgical or transcatheter) at Rigshospitalet, Denmark will be included. Participants will undergo CMR before surgery and at a 1-year follow-up. Other assessments include clinical evaluation and blood sampling. The primary end-point is change in T1 values after AVR.

Hypotheses and perspectives: The investigators hypothesize that (1) myocardial fibrosis* will regress in patients undergoing AVR as a group, (2) the degree of myocardial fibrosis is positively correlated with the degree of symptoms, (3) the regression of myocardial fibrosis is greater in patients undergoing TAVR compared to SAVR, and (4) the regression of myocardial fibrosis is greater in patients with tricuspid aortic stenosis compared to bicuspid aortic stenosis. Ultimately, T1 mapping is a potential marker for improved patient selection for the timing of AVR.

* Estimated by T1 mapping

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Severe aortic valve stenosis (Vmax > 4 m/s and/or mean gradient >40 mmHg)

Exclusion Criteria:

* Reduced left ventricular ejection fraction (<50%)
* More than mild left-sided valvular insufficiency
* Previous or planned primary coronary intervention (PCI) or coronary artery by-pass grafting (CABG)
* Persistent atrial fibrillation
* Contraindications for CMR (pregnancy, severe claustrophobia, magnetic metallic implants)
* Pacemaker/ICD

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from Righospitalet, Denmark, when referred to AVR.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in T1 values from baseline to follow-up | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
New York Heart Association (NYHA) Classification | Through study completion, an average of 1 year
Type of AVR | Through study completion, an average of 1 year
  SAVR or TAVR
Native valve | Through study completion, an average of 1 year
  Bicuspid or tricuspid aortic valve
Left ventricular volumes | Through study completion, an average of 1 year
  By cardiac magnetic resonance
Left ventricular mass | Through study completion, an average of 1 year
  By cardiac magnetic resonance
Left ventricular strain | Through study completion, an average of 1 year
  By cardiac magnetic resonance and echocardiography
Late gadolinium enhancement | Through study completion, an average of 1 year
  By cardiac magnetic resonance
Extracellular volume | Through study completion, an average of 1 year
  By cardiac magnetic resonance
Left ventricular ejection fraction | Through study completion, an average of 1 year
  By cardiac magnetic resonance and echocardiography
Left atrial size | Through study completion, an average of 1 year
  By cardiac magnetic resonance and echocardiography
e' velocity | Through study completion, an average of 1 year
  By echocardiography
E/e' ratio | Through study completion, an average of 1 year
  By echocardiography
Tricuspid regurgitation velocity | Through study completion, an average of 1 year
  By echocardiography
Concentration of NT-Pro-BNP | Through study completion, an average of 1 year
Concentration of Troponin T | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen O, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data can be provided upon request
Time Frame: From study end
Access Criteria: Researchers who provide a methodological sound proposal